CLINICAL TRIAL: NCT01398891
Title: Development of a Positive Psychology Intervention to Reduce Suicide Risk
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Blake 11, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P002826
Record Dates: First submitted 2011-07-15; First posted 2011-07-21 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Suicidal Ideation; Suicide Attempt
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Psychology Exercises (Experimental)
  Interventions: Other: Positive Psychology Exercises

INTERVENTIONS:
Other: Positive Psychology Exercises — At each session, the interventionalist will prepare the subject to complete a randomly-selected positive psychology exercise, lasting approximately 20 minutes, within the next 24 hours. He or she will describe the rationale for the exercise and the details of the exercise, and will answer any questions. A sheet with written instructions (matching the verbal instructions) for the exercise will be provided, with space for recording the exercise and an area to provide ratings on the exercise. On the following day, the interventionalist will review the prior day's exercise (and record whether it was completed). The exercises will be completed daily on weekdays for a maximum of 8 days.

SUMMARY:
This pilot study will recruit patients admitted to the inpatient psychiatric unit at MGH for suicidal ideation or a suicide attempt. Inclusion criteria will be broad to increase enrollment rates and obtain information for patients with a wide range of diagnoses and illness severity. Enrolled subjects will complete randomly-selected positive psychology exercises daily (on weekdays) until discharge and will rate the exercises in multiple domains. Subjects' participation will be complete at the end of their admission or when all exercises have been completed, whichever comes first.

Overall, our goal is to assess the acceptability and utility of eight possible positive psychology interventions related to gratitude, optimism, kindness, mindfulness, recollection, and forgiveness in suicidal inpatients.

This is a single-arm study, completed with patients who have been admitted to the hospital for suicidal ideation or a suicide attempt. It is aimed at developing a positive psychology treatment aimed at suicidal patients. The study consists of serial completion of different positive psychology exercises, once daily, during admission, to get subjects' input on their feasibility and impact. This will allow us to work collaboratively to identify the specific exercises that best fit this population. Subjects' participation ends when they are discharged from the hospital. The investigators plan to enroll 30 subjects at MGH (and total) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older) admitted to inpatient psychiatric unit at Massachusetts General Hospital
* Suicidal ideation at time of admission OR
* Admission occurring in context of suicide attempt
* Ability to read and write in English

Exclusion Criteria:

* Psychotic symptoms
* Cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Completion of exercises | Every 24 hours until all exercises administered or discharge occurs
  Exercises assigned each day and assessed for completion the next day (a total of eight exercises)

SECONDARY OUTCOMES:
Optimism | Baseline and on the date of discharge (average length of admission= 2 weeks)
  Life Orientation Test-Revised
Feasibility and utility of exercises | Assessed within 24 hours of exercise completion
  Self-report using Likert scale
Hopelessness | Baseline and on the date of discharge (average length of admission=2 weeks)
  Beck Hopelessness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States